CLINICAL TRIAL: NCT04927000
Title: The Role of Tofacitinib in Steroid Withdrawal in Rheumatoid Arthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-388
Record Dates: First submitted 2021-05-31; First posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2020-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; tofacitinib; dsease remission
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): All subjects used one or two the basic DMARDs: Methotrexate (10mg) combined with sulfasalazine (2G / day), Iguratimod (50 mg / day), leflunomide (20 mg / day)].
  All subjects were treated with Glucocorticoid (10-15mg)/Days).
- Tofacitinib treatment group (Experimental): All subjects used one or two the basic DMARDs: Methotrexate (10mg) combined with sulfasalazine (2G / day), Iguratimod (50 mg / day), leflunomide (20 mg / day)].
  All subjects were treated with Glucocorticoid (10-15mg)/Days). All subjects were treated with Tofacitinib 5mg/BID.
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — in tofacitinib treatment group，we added tofacitinib 5mg/BID in the basic treatment in all subjects.
  Other Names: Xeljanz
  Arms: Tofacitinib treatment group

SUMMARY:
Rheumatoid arthritis (RA) is a systemic chronic arthritis characterized by systemic inflammation, persistent synovitis and final joint destruction Inflammatory diseases can lead to decreased productivity and impaired health-related quality of life. As a chronic disease, rheumatoid Chronic arthritis needs long-term treatment. At the same time, RA can cause skin, eye, lung, liver, kidney, blood and cardiovascular diseases All of them were extraarticular lesions. It causes a heavy burden to the patients themselves, their families and the society. The main clinical manifestations of RA were morning stiffness Joint swelling and pain, cartilage destruction and joint space narrowing, if not treated, will lead to joint destruction, deformity and dysfunction The rate of disability is high. As a new drug in the treatment of RA, tofacitinib can relieve RA symptoms and promote joint healing It can recover the injury and correct the abnormal immune function. At present, studies have proved that the traditional anti rheumatic drugs are ineffective in the treatment of RA. The addition of tofacitinib to patients may be beneficial to the treatment.

DETAILED DESCRIPTION:
Participant inclusion and selection criteria: A total of 170 patients with rheumatoid arthritis were enrolled.

Inclusion criteria: The diagnosis of rheumatoid arthritis of patients must meet the ACR 1987 classification criteria for rheumatoid arthritis, female, aged 30-65 years old, all The patients have been using traditional dMARDs combined with glucocorticoid for 1 month (glucocorticoid dosage 10-15mg/day), and the DAS28 scores are all greater than 3.2, considering that the disease is still active.

Exclusion criteria: Including other connective tissue diseases, neurological diseases, combined depression, ongoing antidepressant treatment, severe cardiovascular disease, latent tuberculosis, tumors, severe liver and kidney dysfunction.

Randomly divided into two groups: tofacitinib treatment group and control group with 85 cases each. The probability of patients being classified into different groups: both are 50%.

Control group: basic dMARDs of all subjects: methotrexate (10mg) combined with [(sulfasalazine (2g/day), isilamod (50mg/day), leflunomide (20mg/day)] One or two of the two. All subjects used glucocorticoids (10-15 mg/day).

Tofacitinib group: combined with tofacitinib 5mg/twice a day on the basis of the above scheme.

All patients will be evaluated once a month for the first three months, including the DAS28 score, serum C-reactive protein, erythrocyte sedimentation rate, liver and kidney function and other serological indicators. After three months, the disease will be evaluated once 1-2 months. The assessment content is the same as above. .

Research endpoints: 1. After treatment, the DAS28 score is less than 2.6, considering the disease remission, gradually reduce the dose to stop the hormone. 2. Hormone use for more than 6 months cannot be reduced or stopped or if the condition worsens, consider adding other dMARDs or biological agents to control the condition. 3. The test needs to be terminated in case of serious adverse reactions. All subjects recorded the time when hormones were stopped and the total amount of hormones used.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of rheumatoid arthritis female gender, 30 to 65 years old, all patients the traditional DMARDs combined with glucocorticoid for 1 month (glucocorticoid dosage 10-15mg/ day) was used, and DAS28 score was large than 3.2, consider that the disease is still active.

Exclusion Criteria:

other connective tissue diseases, neurological diseases, major depression, cardiovascular disease, latent tuberculosis, tumor, severe liver and kidney dysfunction.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-05-31 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Disease remission of rheumatoid arthritis patients | through study completion，an average of 1 year
  Disease Activity Score 28 score(DAS28). DAS28>3.2 means disease active，DAS28 <2.6 means disease remission
Disease remission of rheumatoid arthritis patients | through study completion，an average of 1 year
  Liver and kidney function were measured with a BN ProSpec System. Alanine aminotransferase more than three times of the normal value and eGRF<60 were exclued for further study.

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China